CLINICAL TRIAL: NCT06408805
Title: Hereditary Angioedema Due to C1 Inhibitor Deficiency: Evaluation of the Cardiac Autonomic Nervous System Profile in Patients With and Without Prophylactic Treatment
Brief Title: Autonomic Nervous System Profile in Hereditary Angioedema
Acronym: ANS-HAE
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 2746CE
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; Heart Rate Variability; Autonomic Nervous System; Rare disease
MeSH Terms: conditions — Angioedemas, Hereditary; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hereditary angioedema: Patients with documented diagnosis of hereditary angioedema due to C1 inhibitor deficiency with or without prophylactic treatment and aged between 18 and 65 years.
- Healthy individuals: Healthy individuals with an age between 18 and 65 and matched with patients with hereditary angioedema by age and gender.

SUMMARY:
The goal of this study is to compare the autonomic nervous system control of patients with hereditary angioedema to healthy individuals.

The main questions it aims to answer are:

Are there differences in the autonomic nervous system control between patients with hereditary angioedema and healthy individuals during short-term resting period and during orthostatic challenges?

Are there differences in the autonomic nervous system control recorded over long-term periods (i.e. 24 hours)?

DETAILED DESCRIPTION:
Angioedema (AE) without wheals is a localized self-limiting edema associated with different mechanisms. The best-known form is hereditary angioedema (HAE) due to C1 inhibitor deficiency (C1-INH), a rare disease with a prevalence of 1:65000 in Italy. Symptoms include swelling of the extremities, genitals, bowel mucosa, face, and upper airway including the larynx. Laryngeal attacks, if not treated, can lead to death. AE attacks are unpredictable and occur episodically upon release of the main mediator of the attack, namely bradykinin, resulting from hyperactivation of the contact system lacking its main control protein C1-INH.

The overall result is an impairment of the endothelial function associated with increased vascular permeability. The release of bradykinin occurs locally, in an unpredictable way, at times facilitated by trauma and different triggers such as stress.

In C1-INH-HAE patients, the autonomic nervous system (ANS) has a role in the regulation of vascular permeability, for example via the baroreflex mechanism. It is also known that sympathetic nervous system inhibition by the α2 agonist clonidine reduces microvascular permeability in endotoxemic animals, suggesting that antagonizing the sympathetic nervous system might prove beneficial in stabilizing capillary leakage during inflammation. Similarly, the vagus nerve has a protective role in models of inflammation such as ischemia-reperfusion injury. The parasympathetic tone, acting on the B2-receptors in the nucleus ambiguous, can also be modulated by bradykinin. The ANS could be investigated using the tilt test and Holter ECG monitoring in current clinical practice when its impairment is suspected. Power spectral analysis of heart rate variability (HRV), i.e. the analysis of the spontaneous fluctuations of the heart period, is exploited to analyze data collected during the tilt test and Holter-ECG, deriving indices of the autonomic control.

In C1-INH-HAE patients the cardiac ANS was investigated during a remission period, during the AE attack and its prodromal phase.

It has been demonstrated that HRV analysis, extended to multiday ECG recordings, may furnish an early marker of an angioedema attack.

In this perspective, the identification of markers, like HRV parameters, could play a crucial role in helping patients and physicians to characterize the ANS control in each patient and individualize treatment based on the ANS balance.

This study aims to compare the cardiovascular ANS control in healthy subjects and HAE patients by head-up tilt test monitoring and evaluate the differences in long-term ANS between healthy controls and HAE patients by Holter ECG monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of hereditary angioedema due to C1 inhibitor deficiency (for the group of patients only)

Exclusion Criteria:

* Any type of chronic diseases requiring chronic treatment.
* Active acute disease
* Sars-Cov2 infection in the previous three months
* Acute attacks experiences within the previous week and within 72 hours after the enrollment
* Patients in prophylaxis treated off-label.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The group of patients with hereditary angioedema were recruited during a out-patient visit in a tertiary care center. The group of healthy individuals were volunteers recruited from community.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Short-term heart rate variability | Baseline
  Changes in heart rate variability indices analyzed during tilt test

SECONDARY OUTCOMES:
Long-term heart rate variability | Baseline
  Changes in heart rate variability indices analyzed during holter ECG recordings
Concentration of catecholamines | Baseline
  Changes in the concentration of catecholamines, quantified in the blood plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Milan, Italy

REFERENCES:
- [Derived] De Maria B, Ranucci L, Gino C, Zulueta A, Parati M, Cesoni Marcelli A, Zingale LC, Sideri R, Dalla Vecchia LA, Perego F. Cardiac and vascular autonomic control in patients with hereditary angioedema. Front Physiol. 2025 Dec 16;16:1690915. doi: 10.3389/fphys.2025.1690915. eCollection 2025. PMID 41476578